CLINICAL TRIAL: NCT03390959
Title: Effectiveness of Proprioceptive Training on Plantar Pressure, Postural Balance, Posture and Gait in Individuals With Diabetes Mellitus Type 2
Brief Title: Effectiveness of Proprioceptive Training on Plantar Pressure, Balance, Posture and Gait in Individuals With Diabetes Mellitus Type 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kelly Antunes e Silva Oliveira (Other)
Responsible Party: Sponsor-Investigator, Kelly Antunes e Silva Oliveira, Bachelor, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Proprioceptive DM2; Feedback N.2.052.913 (Other: UFPE CAAE N. 61248216.2.0000.5208)
Record Dates: First submitted 2017-12-28; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Proprioception; Diabetes Mellitus, Type 2; Postural Balance; Gait; Posture
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two groups: Control Group (CG) and the Trained Group (TG)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor) The one who assess the patients in the beginning and in the final moment (investigator) not know in what group the patient is. As the investigator that will do the statistic (outcome assessor).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Training (Experimental): The group participates in proprioceptive training that promotes sensory integration.
  Interventions: Other: Proprioceptive Training
- Control Group (Other): The group continues in their daily lives with phone monitoring.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Proprioceptive Training — Individuals in the Trained Group will perform the training twice a week for 45 minutes and perform for a period of 12 weeks.
  The training is divided into a pre-training phase where general hip dissociation exercises and simple stretching of the hip flexor and extensor muscle groups, knee, foot and paravertebral are performed.
  The second phase is the proprioceptive training, where it will involve training of balance, sensitivity and proprioception, being used a circuit composed of 15 stations, whose time of stay in each station is 2 minutes.
  And finally the third stage are relaxation exercises, performed with breathing exercises associated with slow active movements of the joints.
  Other Names: Experimental
  Arms: Proprioceptive Training
Other: Control Group — Will not be submitted to any physical intervention. It continues in your daily life with only phone monitoring.
  Arms: Control Group

SUMMARY:
Introduction: Diabetes mellitus (DM) can be considered as one of the most important chronic diseases in the public health system, presenting a high cost for health services. Along with the increase in diagnosed cases of DM, there is a simultaneous increase in DM-related manifestations, such as peripheral diabetic neuropathy, diabetic foot ulcers and amputations. Decreased plantar sensitivity caused by microvascular complications, reduced sensation of vibration and loss of pressure sensitivity may be associated with recurrent falls due to reduced proprioceptive feedback. Although much is known about the beneficial results of physical exercise on glucose metabolism and insulin action, there are still few studies that evaluate the effects of different types of physical exercise, especially proprioceptive training, on plantar pressure, balance and posture of individuals.

Objective: The present study aims to evaluate the efficacy of proprioceptive training on plantar pressure, postural balance and posture in adults with Type 2 Diabetes Mellitus.

Methods: This study is a randomized, double blind, controlled clinical trial (evaluator and statistician) with individuals of both sexes, with type 2 diabetes mellitus diagnosed for at least 3 years, over 45 years of age, that can walk without assistance or supervision of others. Two groups will be formed, the Control Group (CG) and the Trained Group (TG), and the ideal "n" will be calculated in a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* individuals with type 2 diabetes mellitus, diagnosed for at least 3 years
* both genders
* aged 45 years or over
* able to wander without assistance or supervision from others
* absence of macroangiopathy
* no history of neurological, muscular or rheumatic diseases for the etiology of diabetes
* agree to participate in the study, signing the Free and Informed Consent Term (TCLE) pursuant to Resolution 466/12 of the National Health Council

Exclusion Criteria:

* presence of uncontrolled hypertension (systolic ≥ 200 mmHg and / or diastolic ≤100 mmHg);
* presence of a rheumatic condition that makes it impossible to perform the movements performed in the evaluation and in the therapeutic intervention;
* lack of more than 15% to the proprioceptive training program;
* individuals who perform some physical activity
* dependence on alcohol and illicit drugs

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Plantar Pressure | 5 minutes
  Modular baropodometric platform MPS (M.P.S. Loran, KINETEC), where plantar pressure variables are provided in (Kgf / cm²) and plantar surface area (cm²) provided by BIOMECH STUDIO software.
Balance | 5 minutes
  Modular baropodometric platform MPS (M.P.S. Loran, KINETEC), where distance of C.O.P are provide in (mm) and average speed in (mm / sec), provided by BIOMECH STUDIO software.
Posture | 1 hour
  Optoelectronic system (SMART DX100, produced by BTS Bioengineering, Milan, Italy)
Gait | 10 minutes
  The Time Up And Go Test (TUG) was performed using the Wiva® Science sensor KINETEC® type inertial sensor

SECONDARY OUTCOMES:
Plantar Sensitivity | 10 minutes
  The tactile sensitivity will be evaluated in 4 plantar areas: medial forefoot, lateral forefoot, midfoot and hallux, using Semmes-Weinstein (10g) nylon monofilament (SORRI Bauru®).
  Test tubes containing cold and hot water for thermal sensitivity assessment and a clinical tuning for evaluation of vibration sensitivity will also be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Maria das Graças Araujo, Recife, Pernambuco, Brazil